CLINICAL TRIAL: NCT05651633
Title: Effectiveness of Analgesic Ear Drops as add-on Treatment to Oral Analgesics in Children With Acute Otitis Media: a Pragmatic Randomised Controlled Trial
Brief Title: Analgesic Ear Drops for Children With Acute Otitis Media
Acronym: OPTIMA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial accrual problems
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Roderick P. Venekamp, Associate Professor, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80-87200-98-1017; NL9500 (Registry Identifier: Netherlands Trial Register); 10060011910003 (Other Grant/Funding Number: The Netherlands Organisation for Health Research and Development (ZonMw)); 2021-003019-24 (EudraCT Number)
Record Dates: First submitted 2022-11-09; First posted 2022-12-15 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Acute Otitis Media; Pain
MeSH Terms: conditions — Otitis Media; Pain | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: pragmatic, two arm, individually randomised, open, superiority trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine ear drops with usual care (Experimental): usual care: oral analgesic with/without antibiotics
  Interventions: Drug: lidocaine hydrochloride 5mg/g
- usual care (No Intervention): usual care: oral analgesic with/without antibiotics

INTERVENTIONS:
Drug: lidocaine hydrochloride 5mg/g — 1-2 drops up to six times daily for a maximum of 7 days
  Other Names: Otalgan
  Arms: Lidocaine ear drops with usual care

SUMMARY:
This trial aims to investigate whether analgesic ear drops added to usual care provide superior ear pain relief over usual care alone in children presenting to primary care with AOM. Children will be randomly allocated (ratio 1:1) to either 1) lidocaine hydrochloride 5mg/g ear drops (Otalgan) 1-2 drops up to six times daily for a maximum of 7 days in addition to usual care (oral analgesics, with/without antibiotics) or 2) usual care. Parents will complete a symptom diary for 4 weeks as well as generic and disease-specific quality of life questionnaires at baseline and 4 weeks. The primary outcome is the parent-reported ear pain score (0-10) over the first 3 days.

NOTE:

At the time of publication of the study protocol paper, the investigators were unable to make any amendments to the trial registration record in the Netherlands Trial Register (NTR) (NL9500; date of registration: 28 May 2021). The addition of a data sharing plan was required to adhere to the International Committee of Medical Journal Editors (ICMJE) guidelines. The investigators therefore re-registered the trial in ClinicalTrials.gov. This second registration is for modification purposes only and the NTR record (NL9500) should be regarded as the primary trial registration.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 to 6 years
* Parent-reported ear pain in 24 hours prior to enrolment
* GP-diagnosis of (uni- or bilateral) AOM

Exclusion Criteria:

* with (suspected) tympanic membrane perforation or ventilation tubes
* with ear wax obscuring visualisation of the tympanic membrane
* who are systemically very unwell or require hospital admission (e.g. child has signs and symptoms of serious illness and/or complications such as mastoiditis/meningitis)
* who are at high risk of serious complications including children with known immunodeficiency other than partial IgA or IgG2 deficiencies, craniofacial malformation including cleft palate, Down syndrome and previous ear surgery (with the exception of ventilation tubes in the past)
* who have a known allergy or sensitivity to study medication or similar substances (e.g. other amide-type anaesthetics: bupivacaine, mepivacaine, prilocaine, etc)
* who have taken part in any research involving medicines within the last 90 days, or any other AOM-related research within the last 30 days
* who suffer from chronic recurrent pain of another origin than the ear
* who have participated in this trial during prior AOM episode

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2023-12-16 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
The parent-reported ear pain score over the first three days | 3 days
  Parents will record their child's ear pain scores during the first three consecutive days using a 0-10 validated numerical rating scale. Higher scores indicate greater severity.

SECONDARY OUTCOMES:
proportion of children consuming antibiotics | in the first 7 days
proportion of children with oral analgesic use | in the first 7 days
overall symptom burden (crying/distress, disturbed sleep, interference with normal activity, appetite, fever and hearing problems) using a 0-6 Likert scale | in the first 7 days
  higher scores indicate greater severity
number of days with ear pain | during follow up (4 weeks)
number of GP reconsultations with/without subsequent antibiotic prescribing | during follow-up (4 weeks)
number of participants with adverse events | during follow-up (4 weeks)
number of participants with complications of AOM | during follow-up (4 weeks)
costs | during follow-up (4 weeks)
  Mean costs per patient will be compared across the randomisation groups
generic quality of life of the child assessed using the 47-item short-form of the Infant Toddler Quality of Life Questionnaire (ITQOL-SF47) | at baseline and at 4 weeks
  The questionnaire consists of 47 items in the following areas: overall health, physical abilities, growth and development, pain, temperament and moods, behavior, general health, parental emotional impact, parental time impact, and family cohesion. Scale for each area: from 0 (worst health) to 100 (best health)
disease-specific quality of life of the child assessed using the Otitis media-6 (OM-6) questionnaire | at baseline and at 4 weeks
  The 6 questions measure Physical Suffering, Hearing Loss, Speech Impairment, Emotional Distress, Activity Limitations, and Caregiver Concerns. Responses for each item were scored from 1 to 7 (1=Not present/no problem; 2=Hardly a problem at all; 3=Somewhat of a problem; 4=Moderate problem; 5=Quite a bit of a problem; 6=Very much of a problem; 7=Extreme problem). A mean score of all six items comprises the OM Total Score. Higher mean scores of all six items indicate greater severity and impact of OM on the child's QOL.
incremental cost-effectiveness ratios; calculated by dividing the estimated differences in costs between groups by the differences in effects observed | during follow-up (4 weeks)
  i.e. the additional cost per additional 1 point reduction in mean ear pain score over the first three days for the analgesic ear drops group versus the usual care group

CONTACTS AND LOCATIONS:
Overall Officials: Roderick Venekamp, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
On completion of the trial, data will be stored for a minimum of 25 years at a central data drive at the Julius Center. The investigators will publish the metadata in the DataverseNL repository and will provide a persistent identifier. The data will be available to researchers who provide a methodologicaly sound proposal to achieve the aims in the approved proposal. Proposals to gain access to the data should be directed to the principle investigator (RPV). Data requestors will need to sign a data sharing agreement.

REFERENCES:
- [Derived] de Sevaux JLH, Damoiseaux RAMJ, Hullegie S, Sanders EAM, de Wit GA, Zuithoff NPA, Yardley L, Anthierens S, Little P, Hay AD, Schilder AGM, Venekamp RP. Effectiveness of analgesic ear drops as add-on treatment to oral analgesics in children with acute otitis media: study protocol of the OPTIMA pragmatic randomised controlled trial. BMJ Open. 2023 Feb 22;13(2):e062071. doi: 10.1136/bmjopen-2022-062071. PMID 36813504